CLINICAL TRIAL: NCT02526719
Title: Nipple Delay Prior to Nipple Sparing Mastectomy: A Pilot RCT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study design changed, no longer a randomized trial design
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UHN14-7891
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: bilateral prophylactic mastectomies; immediate breast reconstruction; nipple sparing; BRCA1 Protein
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Nipple-Sparing Mastectomy (No Intervention): Patients in the control group will receive usual care. The surgical oncologist will perform the NSM and sentinel lymph node biopsy if indicated (active breast cancer or DCIS). We will submit a nipple core biopsy and a 1cm thick biopsy of immediately retro-areolar ductal tissue for permanent section pathology for control patients, and all patients will have the mastectomy specimen submitted for permanent section pathology. Under the same general anaesthesia, the plastic surgeon will perform the IBR (2-stage tissue expander to implant or 1-stage direct to implant). Patients who later have a positive nipple core and retro-areolar biopsy will have a discussion with the surgical oncologist regarding the need for revision breast surgery to excise the NAC, as is current practice.
- Nipple Delay Intervention (Experimental): Patients in the experimental group will have a nipple-delay intervention in addition to usual care. The nipple delay procedure will be performed by the plastic surgeon in the minor clinic procedure room under local anaesthetic 7 - 21 days prior definitive NSM with IBR. The skin flap will be elevated in the plane of the prophylactic mastectomy beneath the NAC. A nipple core biopsy and a 1cm thick biopsy of immediately subareolar ductal tissue will be submitted for permanent section pathology. This approach is consistent with the previous case series of nipple delay for NSM and approved by the multi-disciplinary breast cancer team at our institutions. Patients that have a positive nipple core or sub-areolar biopsy will have the NAC removed at time of definitive mastectomy.
  Interventions: Procedure: Nipple Delay surgery

INTERVENTIONS:
Procedure: Nipple Delay surgery — The nipple delay surgery will be performed by the plastic surgeon as an outpatient procedure in the minor procedure room under local anaesthetic 7 - 21 days prior definitive NSM with IBR. The skin flap will be elevated in the plane of the prophylactic mastectomy beneath the NAC. A nipple core biopsy and a 1cm thick biopsy of immediately subareolar ductal tissue will be submitted for permanent section pathology. This approach is consistent with the previous case series of nipple delay for NSM and has been approved by the multi-disciplinary breast cancer team at our institutions. Patients that have a positive nipple core or sub-areolar biopsy will have the NAC removed at time of definitive mastectomy.
  Arms: Nipple Delay Intervention

SUMMARY:
The goal of nipple-sparing mastectomy (NSM) with immediate breast reconstruction is to reconstruct a breast mound with preservation a patient's natural skin envelope. Preservation of the nipple and areola complex during mastectomy and breast reconstruction is associated with improved quality of life and a better cosmetic result. However, this surgical technique relies on tenuous blood supply to maintain the nipple and areola. Therefore a certain proportion of women will actually lose their preserved nipple-areolar complex due to vascular insufficiency. Furthermore, some women may find out after a nipple-sparing mastectomy that cancer had invaded the nipple-areolar complex, and would require another operation to completely remove the cancer. Despite these devastating complications, there have been no controlled studies to investigate mechanisms to reduce the chance of their occurrence.

Our research study will use a pre-operative minor procedure to enhance blood flow to the nipple-areola complex prior to standard nipple sparing mastectomy among eligible women undergoing mastectomy for breast cancer or risk reduction. A secondary objective is to test how many women actually have active cancer in their nipple at the time of this minor surgical procedure, prior to standard NSM. The investigators hypothesize that our innovative and novel nipple-delay procedure will reduce the risk of loss of the nipple due to vascular insufficiency and may be of benefit to identify the small proportion of women with nipple-areola complex involvement, in order to optimize the ultimate cancer ablation.

For this study the investigators propose to undertake a Pilot RCT as the first step in the evaluation of a delay procedure prior to NSM, and the results will be used to determine the feasibility and inform the optimal design for a definitive RCT. This study question has the potential to set a new standard of care in the management of women seeking NSM for the management of their breast cancer.

DETAILED DESCRIPTION:
The surgical management of breast cancer has evolved over the last few decades, with cancer extirpation becoming less aggressive in parallel with advances in breast reconstruction. Preservation of the nipple-areolar complex (NAC) at time of mastectomy (nipple-sparing mastectomy, NSM), represents a natural progression within reconstructive and surgical oncology to preserve maximum native skin as is oncologically feasible. NSM is associated with improved satisfaction, body image and psychological adjustment. NSM has received increased attention in the lay media, because the ability to preserve the entire breast envelope appeals to patients facing the decision to undergo mastectomy.

Clinician attention regarding NSM has focused on the oncologic implications of the residual breast tissue. Several systematic reviews of prospective and retrospective studies (level II to IV) have concluded that NSM does not impair overall or breast cancer specific survival outcomes compared to skin-sparing mastectomy. This has fostered the adoption of NSM within North America and Europe. The rate of occult NAC involvement ranges from 6 - 30%.

However, the intended purpose of NSM to preserve the NAC may be circumvented if a tenuous sub-dermal blood supply compromises NAC viability. Rates of NAC necrosis are variable, from 0% to nearly 50% of cases 5,6. Few studies explored strategies to prevent this potentially devastating complication. Recent case series employ the use of the surgical delay phenomenon to improve vascular supply and reduce NAC necrosis during NSM 9,10, however this strategy has not been directly compared with standard NSM.

There have been no controlled studies to investigate mechanisms to reduce the chance of potentially devestating complication of NAC necrosis or minimize the clinical impact of occult tumor involvement in the NAC. Because our study is a pilot feasibility study, we have 3 specific rationale to support our design using a pilot study first:

1. : Given lack of evidence to support impaired cancer outcomes, there has been greater interest in NSM within our breast cancer community. Prior to initiating a full trial, it is paramount to determine the extent to which the intervention can be provided as intended.
2. There are a number of well-described challenges to undertaking a RCT of a surgical intervention, and the extent to which women consent to participate, maintain randomized treatment allocation and adhere to study protocol will inform whether this study is feasible at a larger scale. It has not been determined whether candidates for NSM would accept an additional surgical procedure to reduce the risk of NAC necrosis. Lastly, there is the opportunity to identify and revise organization and protocols prior to execution within a full trial.
3. : Given there is wide variation in reported rates of NAC necrosis, it is important to determine the incidence of NAC necrosis within our institutions and use this information to generate and inform sample size calculation. The direction of benefit and preliminary estimates of the effect of the intervention will clarify the choice of primary and secondary outcomes and feasibility for a larger scale study.

The overarching hypothesis driving the main trial is that patients who are allocated to nipple-delay will have a lower rate of NAC necrosis. Additionally we hypothesize may be of benefit to identify the small proportion of women with nipple-areola complex involvement, in order to optimize the ultimate cancer ablation.

Aim 1: To assess treatment fidelity and acceptability to surgeons of the intervention Hypothesis: This pilot RCT will be acceptable to surgeons, and surgeons will adhere to the treatment group (surgical procedure) to which their patient is randomly allocated. Aim 2: To determine feasibility and acceptability to patients of randomization, treatment uptake and retention and data-collection Hypothesis: This pilot RCT will be feasible to implement and acceptable to patients, and the results will inform planning of the main study. Aim 3: To estimate the proportion of patients in the treatment and control groups that develop NAC necrosis (primary outcome) and a preliminary estimate of the effect of the intervention on NAC necrosis (primary outcome), occult cancer and intra-operative NAC perfusion (secondary outcomes). Hypothesis: This pilot study will provide important information regarding treatment effect estimate and variability (standard deviation) that will be used to guide the design and sample size calculation for the main trial. The overarching hypothesis driving the main trial is that patients who are allocated to nipple-delay will have a lower rate of NAC necrosis.

Pilot outcomes: Treatment fidelity and acceptability to surgeons: We will record the proportion of participants who received their randomly allocated treatment assignment to monitor participant adherence to treatment allocation. We will record reasons why any deviation from study protocol occurred (patient or surgeon-driven), and other organizational barriers to meeting usual care (ex: > 21 days between nipple-delay and NSM for experimental-group patients). Feasibility and acceptability of randomization, treatment allocation and data-collection procedures: Patient recruitment and attrition rates will be recorded. We will measure the proportion of participants that generate complete primary and secondary outcome measurements and baseline questionnaires.

Trial outcomes:

Primary outcome: We will compare the proportion of patients in each group that develop NAC necrosis, defined as necrosis requiring local wound care with dressings or surgical debridement. The proportion of patients in each group that develop total (> 75% of NAC) and partial (25 to 75% of NAC) NAC necrosis will be measured at 2 week and 4 weeks after the definitive NSM procedure by the treating plastic surgeon and surgical oncologist, respectively. We will take photographs to provide objective documentation.

Secondary outcomes:

1. The proportion of women in each group who require secondary NAC excision due to positive pathology review after NSM after the retro-areolar and nipple core biopsy during surgical delay (intervention group) or definitive NSM (control group).
2. To include an objective and immediate measure of NAC perfusion, we will compare the mean perfusion score of the NAC between groups using indocyanine green infusion and the SPY Imaging System (Lifecell Corp.) immediately after tissue expander or implant placement and skin closure during the NSM. We will use this as an objective measure of perfusion but will not influence clinical decision making with regards to NAC viability.

For the pilot, this study is significant to generate high-quality evidence-based data and to determine the feasibility to undertake and complete a full-scale RCT. The overarching study has the potential to influence clinical practice and is very contemporary in the management of patients undergoing mastectomy for breast cancer or risk reduction. If nipple-delay is effective in reducing the rate of NAC necrosis, then our proposed intervention has the potential to change clinical practice for surgeons who treat women with breast cancer or at high risk for development. Furthermore, the identification of occult malignancy within the NAC prior to planned NSM may contribute to improved cancer outcomes by not sparing the NAC at the time of mastectomy. We hypothesize a positive outcome would engender support within the breast cancer community to uptake an additional stage. Therefore, our proposed study can be used as a model to incorporate level I evidence into the plastic surgery research community, as well as provide robust data to support a change in clinical practice to improve patient outcomes among women undergoing NSM for breast cancer risk-reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18 years and above
2. Implant-based immediate breast reconstruction
3. Prophylactic mastectomy for risk reduction OR
4. Therapeutic mastectomy for ductal carcinoma in situ (DCIS) or early stage breast cancer where:

a. Tumor size < 3cm b. Tumor to nipple distance > 2cm c. Clinically negative lymph nodes d. No skin involvement, inflammatory breast cancer or Paget's disease

Exclusion Criteria:

1. Previous ipsilateral breast irradiation
2. Regnault ptosis grade II or III
3. Breast size of D cup or greater
4. Active smoker 7. Are there any age,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Nipple-areolar complex (NAC) | NAC necrosis will be measured at 2 week and 4 weeks after the definitive NSM procedure by the treating plastic surgeon and surgical oncologist, respectively.
  We will compare the proportion of patients in each group that develop NAC necrosis, defined as necrosis requiring local wound care with dressings or surgical debridement. The proportion of patients in each group that develop total (> 75% of NAC) and partial (25 to 75% of NAC) NAC necrosis will be measured at 2 week and 4 weeks after the definitive NSM procedure by the treating plastic surgeon and surgical oncologist, respectively. We will take photographs to provide objective documentation.